CLINICAL TRIAL: NCT00336843
Title: Combining 90Y-ibritumomab Tiuxetan With High-dose Chemotherapy of BuCyE and Autologous Stem Cell Transplantation in Patients With B-cell Non-Hodgkin's Lymphoma - an Open-labeled Phase II Study
Brief Title: Zevalin Plus BuCyE High-dose Therapy in B-cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Principal Investigator, Cheolwon Suh, ASCT team, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC 2005-276
Record Dates: First submitted 2006-06-13; First posted 2006-06-14 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Zevalin; B-cell non-Hodgkin's lymphoma; autologous stem cell transplantation; BuCyE regimen
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zevalin-BuCyE (Experimental): histologically confirmed, relapsed or refractory CD20 positive B-cell NHL including diffuse large B-cell, follicular, mantle cell, and Burkitt lymphomas.
  Interventions: Drug: Zevalin-BuCyE

INTERVENTIONS:
Drug: Zevalin-BuCyE — rituximab (IV, 250 mg/m2 on days -21 and -14) single dose of 90Y-ibritumomab (IV, 0.4 mCi/kg on day -14) Busulfan (IV, 0.8 mg/kg every 6 h from day -7 to day -5) Cyclophosphamide (IV, 50 mg/kg on days -3 and -2) Etoposide (IV, 200 mg/m2 every 12 h on days -5 and -4) Autologous stem cells infusion on day 0

SUMMARY:
In order to improve the clinical result of high-dose chemotherapy and autologous stem cell transplantation for B-cell non-Hodgkin's lymphoma, Zevalin will be added to the conditioning regimen. Investigators expect this radioimmunotherapy of Zevalin plus busulfan, cyclophosphamide and etoposide regimen will improve survival of relapsed or poor-risk B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
Title: Combining 90Y-Ibritumomab tiuxetan (Zevalin) with high-dose chemotherapy of BuCyE and autologous stem cell transplantation in patients with relapsed, refractory, or high-risk B-cell non-Hodgkin's lymphoma - an open-labeled phase II study.

Study design: Prospective, multicenter, open-labeled, phase II trial.

Study objectives:

* Primary: event-free survival time following autologous stem cell transplantation with 90Y-Ibritumomab tiuxetan and BuCyE high-dose chemotherapy in patients with relapsed, refractory, or high-risk B-cell non-Hodgkin's lymphoma
* Secondary: overall survival response rate toxicity of the treatment combination

Treatment:

Z-BuCyE Regimen

* Day 21: rituximab, 250 mg/m2, I.V.
* Day 14: rituximab, 250 mg/m2, I.V. 90Y-Ibritumomab tiuxetan, 0.4 mCi/kg, I.V.
* Day 7, 6, 5: busulfan 3.2 mg/kg I.V.
* Day 5, 4: etoposide 200 mg/m2 I.V. every 12 hours
* Day 3, 2: Cytoxan 50 mg/kg I.V.
* Day 0: autologous stem cell infusion

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed B-cell NHL in chemotherapy-sensitive relapse, in partial response to 1st line chemotherapy, or in complete response after 1st line chemotherapy with high IPI score at diagnosis
* Age < 65 years old
* WHO performance status (PS) of 0-2
* ANC > 1,500/mm3, platelet > 100,000/mm3
* Cr < 2.0 mg% or Ccr > 50 mL/min
* Transaminase < 3X upper normal value
* Bilirubin < 2 mg/dL
* Life expectancy of at least 3 months
* Written informed consent
* Optimal harvest of autologous stem cells (CD34+ cells > 5 million/kg plus 2 million/kg for back-up)

Exclusion Criteria:

* Prior hematopoietic stem cell transplantation
* Prior RIT
* Prior external radiation to > 25% of active bone marrow
* CNS involvement of non-Hodgkin's lymphoma
* Serious comorbid diseases
* HIV or HTLV-1 associated malignancy
* History of other malignant disease in the previous 5 years, except squamous cell or basal cell carcinoma of skin or stage I uterine cervical carcinoma or cervical carcinoma in situ
* Known hypersensitivity to murine antibodies/proteins
* Pregnant or breast feeding female patients, adults without effective contraception up to 12 months after RIT
* Persistent toxic side effects from prior therapy
* Prior biologic or immunotherapy less than 4 weeks prior to entry on this study
* Investigational drugs less than 4 weeks prior to entry on this study

Max Age: 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2005-11; Primary Completion 2009-02 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Event-free survival | the time from stem cell infusion to failure or death from any cause
  Three year event-free survival rate would be reported.

SECONDARY OUTCOMES:
Overall survival | from stem cell infusion to death of any cause or last follow-up
  Three year overall survival would be reported.
Toxicity of the treatment combination | any toxicity due to study treatment during study period
  Adverse events would be assessed and graded according to the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE), version 3.0. And the frequency of each grade would be reported as case number and proportion.

CONTACTS AND LOCATIONS:
Overall Officials: Cheolwon Suh, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Departement of Internal Medicine, Division of Oncology, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kang BW, Kim WS, Kim C, Jang G, Lee SS, Choi YH, Lee DH, Kim SW, Kim S, Ryu JS, Huh J, Lee JS, Suh C. Yttrium-90-ibritumomab tiuxetan in combination with intravenous busulfan, cyclophosphamide, and etoposide followed by autologous stem cell transplantation in patients with relapsed or refractory B-cell non-Hodgkin's lymphoma. Invest New Drugs. 2010 Aug;28(4):516-22. doi: 10.1007/s10637-009-9283-z. Epub 2009 Jun 23. PMID 19547918